CLINICAL TRIAL: NCT03446313
Title: A Technology-Based Adaptive Intervention to Promote Cardiovascular Health After Completion of Cardiac Rehabilitation (Mobile4Heart)
Brief Title: Technology-Based Intervention to Promote Heart Health After Cardiac Rehab (Mobile4Heart)
Acronym: Mobile4Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mobile4Heart; 17-22717 (Other: University of California, San Francisco)
Record Dates: First submitted 2018-02-14; First posted 2018-02-26 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Heart Disease; Unstable Angina; Systolic Heart Failure; Cardiovascular Diseases
MeSH Terms: conditions — Myocardial Ischemia; Angina, Unstable; Heart Failure, Systolic; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVN Group (Experimental): Participants assigned to the MVN Group will be using the Movn Rehab mobile app after they are discharged from cardiac rehab.
  Interventions: Behavioral: Movn Mobile App
- Usual Care (No Intervention): Participants assigned to the Usual Care group will receive standard instructions and educational handouts after they are discharged from cardiac rehab.

INTERVENTIONS:
Behavioral: Movn Mobile App — The Movn app will have each participant's personalized instructions for post-cardiac rehab integrated into it including medication reminders, physical activity prompts, educational materials, and patient-reported outcomes.
  Arms: MVN Group

SUMMARY:
The purpose of this study is to determine whether using a mobile app increases adherence to a heart healthy prescription after discharge from a cardiac rehab program.

DETAILED DESCRIPTION:
Ongoing maintenance of physical activity after cardiac rehab is an important part of preventing secondary cardiac events in patients with ischemic heart disease. Our central hypothesis is that monitoring and promotion of health-related behaviors by increasing patient-provider communication through a mobile device after discharge from cardiac rehab increased adherence to a heart healthy prescription over time. Participants will be randomly assigned to use a mobile app or serve as the control group. All participants will have an activity tracker to track their activity for two months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* History of cardiovascular disease that qualified patient for cardiac rehab (i.e. ischemic heart disease, history of unstable angina, systolic heart failure with ejection fraction at 35% or less, and Class II to IV symptoms, coronary artery bypass graft surgery, valve replacement)
* Own a smartphone or tablet

Exclusion Criteria:

* Cognitive impairment
* Lack of English proficiency/literacy
* Clinical conditions including: unstable arrhythmias, aortic stenosis, thrombophlebitis, dissecting aneurysm, symptomatic anemia, active infection, uncontrolled hypertension (resting diastolic > 100 mmHg, systolic > 180 mmHg), decompensated heart failure NYHA class 3-4, current unstable angina, 2nd or 3rd degree heart block, or uncontrolled high grade exercise-induced ventricular ectopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Park, PhD, Principal Investigator — UCSF, John Muir Medical Center
Locations (2):
- United States (2):
  - John Muir Medical Center, Concord, California
  - John Muir Medical Center, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park LG, Elnaggar A, Lee SJ, Merek S, Hoffmann TJ, Von Oppenfeld J, Ignacio N, Whooley MA. Mobile Health Intervention Promoting Physical Activity in Adults Post Cardiac Rehabilitation: Pilot Randomized Controlled Trial. JMIR Form Res. 2021 Apr 16;5(4):e20468. doi: 10.2196/20468. PMID 33861204

RESULTS

PARTICIPANT FLOW:
Groups:
- MVN Group: The intervention group received (1) a Charge 2 (Fitbit Inc) to record step counts, (2) a Movn mobile app to record exercise, and (3) push-through motivational PA prompts and educational messages related to CVD management. Messages were sent from the study team through the Movn app as a push notification 3 times per week on random days between 9 AM and 6 PM to provide positive feedback and additional motivation for PA. These 1- and 2-way messages were based on the American Heart Association Simple 7 principles [24] and prompted participants to engage in PA, keep healthy eating habits, or track their medication use.
  Additionally, participants could use the Movn app to record daily weight, blood pressure, heart rate, medication use, and other exercise (eg, swimming, biking) not captured by the Fitbit device. Every time they chose to record any of these other measures, they were prompted to complete this information through a push notification from the app. Finally, mHealth participants had the ability to report any cardiovascular symptoms through the Movn app. If the participant reported shortness of breath or chest pain, a message prompted them with a button to call 911. The study team triaged participant entries once a day.
- Usual Care: Participants in the control group were provided a basic pedometer (Walking 3D, IceFox) and paper-and-pencil diary to record daily step counts. They were asked to fasten the pedometer around their waist or to place it in their pants pocket during all waking hours.
  All participants received a phone call (or text message if in the intervention group) 3 days following enrollment to answer any questions regarding the study and verify adherence to the assigned regimen. After 1 month of participation, participants received a follow-up phone call or text sent by the study staff.
Period: Overall Study
Arm/Group | MVN Group | Usual Care
Started | 32 | 28
Completed | 26 | 25
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Failed primary screening | 3 | 0
Not completed — Diagnosed with terminal cancer | 1 | 0
Not completed — Excluded from analysis | 1 | 1

BASELINE CHARACTERISTICS:
Population: We enrolled 60 individuals; however, 9 withdrew or were lost to follow-up (6 from the intervention group and 3 from the control group), representing 15% (9/60) attrition.
Groups:
- Total: Total of all reporting groups
Arm/Group | MVN Group | Usual Care | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants] — Population: We enrolled 60 individuals; however, 9 withdrew or were lost to follow-up (6 from the intervention group and 3 from the control group), representing 15% (9/60) attrition.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 11 | 11 | 22
    >=65 years | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.6) | 66.8 (8.7) | 66.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 22 | 41
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Steps Per Day
Description: Physical activity will be measured by steps per day using activity tracker.
Time Frame: Two months
Measure: Mean (Standard Deviation); unit: Steps/day
Arm/Group | MVN Group | Usual Care
Number analyzed (Participants) | 26 | 25
Steps/day | 8860 (5334) | 6633 (4684)

2. Primary Outcome: 6MWT
Description: Physical activity will be measured by a six minute walk test.
Time Frame: 2 months
Measure: Mean (Standard Error); unit: meters
Arm/Group | MVN Group | Usual Care
Number analyzed (Participants) | 26 | 25
meters | 430 (112) | 429 (97)

3. Secondary Outcome: PHQ-9
Description: Depression will be measured by the Patient Health Questionnaire-9 (PHQ-9). Scores range from 0 (lowest) to 27 (highest), higher score associated with moderate to severe depression.
Time Frame: 2 months
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Groups:
- MOVN: The intervention group received (1) a Charge 2 (Fitbit Inc) to record step counts, (2) a Movn mobile app to record exercise, and (3) push-through motivational PA prompts and educational messages related to CVD management. Messages were sent from the study team through the Movn app as a push notification 3 times per week on random days between 9 AM and 6 PM to provide positive feedback and additional motivation for PA. These 1- and 2-way messages were based on the American Heart Association Simple 7 principles [24] and prompted participants to engage in PA, keep healthy eating habits, or track their medication use.
  Additionally, participants could use the Movn app to record daily weight, blood pressure, heart rate, medication use, and other exercise (eg, swimming, biking) not captured by the Fitbit device. Every time they chose to record any of these other measures, they were prompted to complete this information through a push notification from the app. Finally, mHealth participants had the ability to report any cardiovascular symptoms through the Movn app. If the participant reported shortness of breath or chest pain, a message prompted them with a button to call 911. The study team triaged participant entries once a day.
- Usual Care: Participants in the control group were provided a basic pedometer (Walking 3D, IceFox) and paper-and-pencil diary to record daily step counts. They were asked to fasten the pedometer around their waist or to place it in their pants pocket during all waking hours.
Arm/Group | MOVN | Usual Care
Number analyzed (Participants) | 26 | 25
score on a scale | 1 [0 to 3] | 2 [0 to 3]

4. Secondary Outcome: Exercise Self-Efficacy Scale (EXSE)
Description: Self-efficacy will be measured by the Exercise Self-Efficacy Scale (EXSE). Scores can range from 0 (lowest) to 100 (highest) with 0 indicating low self-efficacy and 100 indicating high self-efficacy.
Time Frame: 2 months
Population: Total scores for depressive symptoms and exercise self-efficacy were examined from baseline to 2 months. We also examined these variables as possible covariates related to the PA and 6MWT results.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | MVN Group | Usual Care
Number analyzed (Participants) | 26 | 25
score on a scale | 10 [9.9 to 10] | 9.9 [8.4 to 10]

5. Secondary Outcome: Acceptability
Description: Satification survey, scored 0 (lowest) to 5 (highest), higher score associated with greater satisfaction
Time Frame: 2 months
Population: Surveys were given to participants in the intervention group who agreed to participate in individual interviews.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MVN Group | Usual Care
Number analyzed (Participants) | 7 | 0
Score on a scale
  Fitbit device | 4.83 (0.41) |
  Movn app | 4.5 (0.71) |

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | MVN Group | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/28
Other Adverse Events (participants affected / at risk) | 0/32 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVN Group (N=32) | Usual Care (N=28)
Terminal cancer diagnosis unrelated to study (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03446313/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03446313/SAP_001.pdf